CLINICAL TRIAL: NCT06641583
Title: Efficacy of LEGO Therapy for Adolescent with Level 1 Autism
Acronym: LEGO
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Narzisi (Other)
Responsible Party: Sponsor-Investigator, Antonio Narzisi, PhD, IRCCS Fondazione Stella Maris
Organization: IRCCS Fondazione Stella Maris (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: LEGO 126/2024
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Neurodevelopmental Disorder
Keywords: Autism Spectrum Disorder; ADHD
MeSH Terms: conditions — Neurodevelopmental Disorders; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exprimental (Experimental): Experimental Group: This group will consist of children aged 10-14 diagnosed with high-functioning Autism Spectrum Disorder (ASD). These children will participate in LEGO therapy sessions once a week for 90 minutes over the course of 3 months (12 sessions total). The goal is to evaluate how LEGO therapy influences their social skills and behavior.
  Interventions: Behavioral: LEGO
- Control (Active Comparator): Control Group: This group will also consist of children aged 10-14 diagnosed with high-functioning ASD. However, these children will not receive LEGO therapy. Instead, they will continue their usual treatments in their local settings without participating in the LEGO therapy sessions. This group's outcomes will be compared with the experimental group to assess the effectiveness of LEGO therapy.
  Interventions: Other: Controllo

INTERVENTIONS:
Behavioral: LEGO — The LEGO Therapy intervention in this clinical trial is designed to enhance social skills in children with high-functioning Autism Spectrum Disorder (ASD). The intervention involves the following components:
  Group Sessions: The therapy will be conducted in small groups of three children of the same age (10-14 years) with a diagnosis of high-functioning ASD. The sessions are designed to foster collaboration and social interaction between the participants.
  Duration: The intervention will last for 3 months, consisting of 12 sessions, with each session lasting 90 minutes. Sessions will take place once a week at the IRCCS Fondazione Stella Maris.
  Supervision: The groups will be supervised by trained professionals specializing in neurodevelopmental disorders, ensuring that the therapy is structured and supportive of each child&#39;s individual needs.
  Therapy Structure: During the sessions, children will engage in LEGO-based tasks, where they collaborate to build LEGO models.
  Arms: Exprimental
Other: Controllo — This group will also consist of children aged 10-14 diagnosed with high-functioning ASD. However, these children will not receive LEGO therapy. Instead, they will continue their usual treatments in their local settings without participating in the LEGO therapy sessions. This group's outcomes will be compared with the experimental group to assess the effectiveness of LEGO therapy.
  Arms: Control

SUMMARY:
The goal of this clinical trial is to learn if LEGO therapy can enhance social skills in children aged 10-14 diagnosed with high-functioning Autism Spectrum Disorder. The main questions it aims to answer are:

Does LEGO therapy improve social communication and interaction skills in children with Autism Spectrum Disorder? Do children show behavioral improvements in social skills after participating in LEGO therapy? Researchers will compare children receiving LEGO therapy to a control group (who will not receive LEGO therapy but continue their usual treatments) to see if LEGO therapy leads to greater improvements in social skills.

Participants will:

Complete behavioral tasks, including a LEGO construction test, at the beginning (T0) and after 3 months (T1).

Attend weekly LEGO therapy sessions for 90 minutes, over the course of 3 months (12 sessions).

Complete questionnaires about social behaviors, both parents and children, at T0 and T1.

DETAILED DESCRIPTION:
The study aims to involve children with Autism in a social skills enhancement program called LEGO therapy. The program will consist of 12 sessions (over 3 months), held once a week for 90 minutes. These sessions will take place at the IRCCS Fondazione Stella Maris in Calambrone (Pisa). Before the program starts (T0) and after it ends (T1, 3 months later), both parents and their children will be asked to complete some questionnaires designed to investigate potential changes in certain behavioral variables before and after the LEGO Therapy intervention. Additionally, at both T0 and T1, children will also be assessed through a LEGO construction task.

LEGO Therapy Intervention The LEGO therapy sessions will be conducted in a group setting. The group will consist of three children of the same age, all diagnosed with high-functioning Autism Spectrum Disorder. The group will be supervised by staff specialized in neurodevelopmental disorders. Participation is voluntary, and partecipants may withdraw from the study at any time, for any reason, without penalty. All collected data will remain anonymous and analyzed in aggregate form. The questionnaires are not designed to collect personal information about parents or their children. The study does not intend to evaluate other aspects beyond those specified, and no incidental findings (e.g., clinical or diagnostic) are expected. The collected data will be stored on a private server and only accessible to the study supervisors (i.e., not provided to third parties) for five years. The results will be used for publications and presentations in academic and scientific settings. Participation in the study poses no specific risks, and children can pause and resume the questionnaire at any time. If partecipants have any questions or concerns about the nature of this research, please contact the lead researcher Antonio Narzisi at IRCCS Fondazione Stella Maris, 050886308, antonio.narzisi@fsm.unipi.it.

What are the characteristics of this study?

This is an interventional study involving 64 subjects with Autism Spectrum Disorder (both male and female), aged 10 to 14. The children will be consecutively recruited either from natural admissions to the IRCCS Fondazione Stella Maris - Operational Unit 2 of Child and Adolescent Psychiatry and Psychopharmacology or through outpatient services. The study will last 6 months, during which time the investigators plan to engage participants. Specifically, this is an open-label randomized study, meaning that both the experimenter and the participant will know the type of treatment being studied. The investigators recognize that open-label studies can introduce bias due to participants and caregivers being aware of the treatment. However, the investigators are implementing several strategies to mitigate these biases:

Blinding of Assessors: The outcome assessors will be unaware of the treatment group to which the participants have been assigned, reducing the risk of bias in outcome assessments.

Use of Objective Measures: The investigators will include objective and standardized measures to evaluate outcomes, in addition to subjective assessments from participants and caregivers.

Data Analysis: The investigators will perform rigorous statistical analyses to control for and identify potential confounding effects related to treatment awareness.

Even though LEGO therapy is well-structured and has demonstrated efficacy in the United States, the investigators cannot assume that the results will automatically translate to the Italian context. Cultural, social, and systemic differences may influence treatment effectiveness. Therefore, a local evaluation of effectiveness is essential to:

1. Validate the Intervention: Confirm that the therapy produces the same benefits in the new cultural context.
2. Adapt the Protocol: Identify and make any necessary adjustments to optimize the intervention for the Italian population.
3. Generate Local Evidence: Provide relevant data for healthcare professionals and policymakers in Italy, supporting the adoption of therapy based on local evidence.

In summary, assessing the effectiveness and cultural adaptability of LEGO therapy in the Italian context is crucial to ensure the treatment is not only applicable but also effective for the new target population. The investigators are aware of the challenges associated with bias in open-label studies and are implementing strategies to mitigate them while ensuring robust and reliable results.

What exams, tests, and procedures are included in the study? If parents decide to allow their child to participate in the study, please note that it involves the administration of certain questionnaires and semi-structured interviews to both parents and their children, as part of routine clinical practice. Specifically, parents will be asked to complete some questionnaires at baseline (T0) and at T1 (after 3 months), with an estimated completion time of around 60 minutes.

Additionally, all children will undergo a behavioral task at both T0 and T1, where they will be engaged in building a LEGO composition on their own and in collaboration with an examiner. The tasks will be recorded and will last no longer than 10 minutes.

After the T0 evaluation, the children will be randomized into two groups: experimental (LEGO therapy) and control (not receiving LEGO therapy). The experimental group will attend weekly LEGO therapy sessions at IRCCS Stella Maris, lasting 90 minutes, for three months (12 sessions). The control group will continue their regular therapies in their local areas and will not receive LEGO therapy. As stated earlier, at the end of the three-month intervention, both experimental and control groups will undergo an outcome assessment, which will take place at IRCCS Stella Maris.

ELIGIBILITY:
Inclusion Criteria:

* age between 10 and 14 years;
* clinical diagnosis of Autism Spectrum Disorder according to ICD-10 (WHO, 1992);
* intellectual level in the normal range (IQ>85);
* self-motivation to participate in the treatment both as regards the adolescent and the family;
* availability of caregiver support the participant during the programme;
* consent of the parents and the adolescent to participate in all evaluations and to be recorded during treatment sessions.

Exclusion Criteria:

* presence of a concomitant major psychiatric disorder (e.g., schizophrenia bipolar disorder);
* presence of oppositional/aggressive behaviour (outside the family context) family context);
* presence of genetic syndromes associated with autism spectrum disorder.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2024-09-20 (Actual); Primary Completion 2025-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Social Skills | From enrollment (T0) to the end of treatment at 12 weeks
  1. Social Skills Improvement System RatingScales (SSiS) (Gresham & Elliott, 2008). The Social Skills Improvement System-Rating Scales (SSIS-RS; Gresham & Elliott, 2008) is a multi-rater (teacher, parent/caregiver, and student) series of rating scales that documents the frequency of social skills and competing problem behaviors. It is a revision of the Social Skills Rating System (SSRS; Gresham & Elliott, 1990). The SSIS-RS assess three domains of social skills, problem behaviors, and academic competence. All forms include common social skills in multiple subdomains: communication, cooperation, assertion, responsibility, empathy, engagement, and self-control. The subscales are grouped beneath Problem Behavior and Social Skills domains. Higher scores mean a better.

SECONDARY OUTCOMES:
Autistic symtoms | From enrollment (T0) to the end of treatment at 12 weeks
  1. ADOS-BOSCC (Lord Group). The brief observation of social communication change (BOSCC) was specifically developed to measure change of core autistic symptoms, for example, for use as outcome measure in early intervention trials. Higher scores mean a worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Cioni, Neurolgy, Study Director — IRCCS Fondazione Stella Maris; Antonio Narzisi, Psychology, Principal Investigator — IRCCS Fondazione Stella Maris
Locations (1):
- Antonio Narzisi, Pisa, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
all IPD collected throughout the trial
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from 01-01-2026 for 5 years
Access Criteria: Writing a mail to principal investigator